CLINICAL TRIAL: NCT00176384
Title: Impact of Three Months of Aerobic Exercise Training on Exercise Capacity and Peripheral Maladaptations in Patients With Severe Chronic Heart Failure (NYHA III b)
Brief Title: Impact of Exercise Training on Exercise Capacity in Patients With Severe Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: F21/02
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Heart Failure
Keywords: chronic heart failure; exercise training
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Behavioral: Aerobic endurance exercise training (ergometer)

SUMMARY:
Patients with heart failure are limited in their exercise capacity due to skeletal muscle alteration and an impairment of peripheral perfusion. Regular physical exercise training has been shown to partially correct these peripheral maladaptations in patients with stable heart failure, which was associated with an improvement in exercise capacity. However, it is unknown so far, whether regular physical activity also exerts beneficial effects in patients with severe chronic heart failure.

Aim of the trial is therefore to assess the effects of aerobic exercise training on exercise capacity, muscle maladaptations and peripheral perfusion in patients with severe chronic heart failure according to NYHA class III b.

DETAILED DESCRIPTION:
A total of 36 patients with severe chronic heart failure are prospectively randomized to either 3 months of aerobic ergometer training or a sedentary control group.

Before and after the intervention period maximal exercise capacity is assessed by ergospirometry, endothelial function is determined by high-resolution A-mode ultrasound, and muscle mass is determined by CT. Skeletal muscle biopsies are obtained at begin and after 3 months and are analyzed for markers of muscle catabolism/anabolism.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure (NYHA class III b)
* peak oxygen uptake <20 mL/min/kg body weight
* left ventricular ejection fraction <25 %
* left ventricular end-diastolic diameter >60 mm

Exclusion Criteria:

* exercise-induced myocardial ischemia
* cardiac decompensation within the last 8 weeks
* ventricular arrhythmias (>Lown 4b) in patients not protected by an ICD
* insulin-dependent diabetes mellitus
* uncontrolled arterial hypertension
* orthopedic conditions excluding training participation
* body mass index >30 kg/m2

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake

SECONDARY OUTCOMES:
Endothelial function
Skeletal muscle mass
Markers of muscle anabolism / catabolism

CONTACTS AND LOCATIONS:
Overall Officials: Rainer P Hambrecht, MD, Principal Investigator — University of Leipzig, Heart Center, Department of Internal Medicine / Cardiology, Leipzig, Germany
Locations (1):
- University of Leipzig, Heart Center, Department of Internal Medicine / Cardiology, Leipzig, Saxony, Germany

REFERENCES:
- [Derived] Erbs S, Hollriegel R, Linke A, Beck EB, Adams V, Gielen S, Mobius-Winkler S, Sandri M, Krankel N, Hambrecht R, Schuler G. Exercise training in patients with advanced chronic heart failure (NYHA IIIb) promotes restoration of peripheral vasomotor function, induction of endogenous regeneration, and improvement of left ventricular function. Circ Heart Fail. 2010 Jul;3(4):486-94. doi: 10.1161/CIRCHEARTFAILURE.109.868992. Epub 2010 Apr 29. PMID 20430934